CLINICAL TRIAL: NCT02614560
Title: A Phase 1/2 Study of Vadastuximab Talirine Administered in Sequence With Allogeneic Hematopoietic Stem Cell Transplant in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study of Vadastuximab Talirine Given Prior to or After Allogeneic Hematopoietic Stem Cell Transplant in AML Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN33A-003
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; AML; antibody-drug conjugate
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Melphalan; vadastuximab talirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-allo (before stem cell transplant) (Experimental): Pre-allo reduced intensity chemotherapy vadastuximab talirine (melphalan and fludarabine)
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: vadastuximab talirine
- Post-allo (after stem cell transplant) (Experimental): Post-allo vadastuximab talirine
  Interventions: Drug: vadastuximab talirine

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2/day intravenously, 5 to 2 days before the transplant (total dose of 120 mg/m2)
  Arms: Pre-allo (before stem cell transplant)
Drug: Melphalan — Melphalan 140 mg/m2 intravenously, 2 days before the transplant
  Arms: Pre-allo (before stem cell transplant)
Drug: vadastuximab talirine — Pre-allo (before stem cell transplant) given 14 days before the stem cell transplant
  Arms: Pre-allo (before stem cell transplant)
Drug: vadastuximab talirine — Post-allo (after stem cell transplant) given on Day 1 of each cycle
  Arms: Post-allo (after stem cell transplant)

SUMMARY:
This study will examine the safety and anti-leukemic profile of SGN-CD33A (vadastuximab talirine) in patients with relapsed chemo-resistant AML, who are given vadastuximab talirine in sequence with standard treatments before a planned stem cell transplant, or as maintenance therapy after a stem cell transplant. The main purpose of the study is to find the best dose and determine the anti-leukemic activity of vadastuximab talirine, given either pre- or post-allogeneic stem cell transplant (alloSCT) for adults with relapsed or refractory AML. This will be determined by assessing the safety and tolerability of vadastuximab talirine. In addition, the pharmacokinetic profile and anti-leukemic activity of the study treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory acute myeloid leukemia (AML) except for acute promyelocytic leukemia
* Eastern Cooperative Oncology Group status of 0 or 1
* Adequate baseline renal and hepatic function
* For Pre-allo Part A (before stem cell transplant): Relapsed or refractory AML (greater than 5% blasts)
* For Pre-allo Part A (before stem cell transplant): Availability of an HLA matched related or unrelated donor
* For Pre-allo Part A (before stem cell transplant): Eligible for an allogeneic hematopoietic stem cell transplant
* For Post-allo Part B: Transplant must have been performed with active AML (greater than 5% blasts) using a conventional conditioning regimen and have achieved CR or CRi post-alloSCT (with ANC greater than or equal to 1,000 and platelet greater than or equal to 50,000)
* For Post-allo Part B: Treatment must begin at least 42 days, but no more than 100 days post-transplant.

Exclusion Criteria:

* Inadequate heart function
* Inadequate lung function
* Previous central nervous system leukemia
* Any history of another metastatic malignancy
* Anti-leukemia treatment within14 days of study drug (other than hydroxyurea or 6-mercaptopurine), immunosuppressive therapy (except for GVHD treatment/prophylaxis in Part B), or investigational agents
* For Pre-allo Part A (before stem cell transplant): Partially matched donors (related or unrelated) and umbilical cord blood cells are excluded as the source of hematopoietic stem cells
* For Pre-allo Part A (before stem cell transplant): Prior alloSCT
* For Post-allo Part B: Active GVHD Grade 2 or higher
* For Post-allo Part B:History of veno-occlusive disease requiring defibrotide
* For Post-allo Part B: History of Grade 2 or higher hepatic GVHD
* For Post-allo Part B: Concurrent use of corticosteroids equivalent of prednisone at a dose of greater than 0.5 mg/kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-10 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Garfin, MD, PhD, Study Director — Seagen Inc.
Locations (11):
- United States (11):
  - City of Hope National Medical Center, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Case Western Reserve University / University Hospitals Case Medical Center, Cleveland, Ohio
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant)
Started | 6 | 8
Completed | 0 | 6
Not Completed | 6 | 2
Not completed — Death | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant) | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Median (Full Range); unit: years] | 58.0 [50 to 69] | 58.0 [25 to 64] | 58.0 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed less than 50% of the time; 3= In bed more than 50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0: Normal activity | 0 | 1 | 1
    Grade 1: Symptoms but ambulatory | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: AE: Adverse events; TEAE: Treatment-emergent adverse event. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), v4.03. Grade 1 = mild, no intervention needed; Grade 2 = moderate, minimal intervention needed; Grade 3 = severe or medically significant, hospitalization is required; Grade 4 = life-threatening, urgent intervention needed; Grade 5 = death related to adverse event. An AE is considered serious if it was fatal, life threatening, required hospitalization, was disabling/incapacitating, resulted in a birth defect or congenital anomally, or was otherwise considered to be medically significant.
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant)
Number analyzed (Participants) | 6 | 8
Participants
  TEAEs | 6 | 8
  AEs Related to Vadatuximab Talirine | 6 | 7
  AEs Leading to Treatment Discontinuation | 0 | 1
  Grade 3 or Higher TEAEs | 6 | 6
  Serious AEs | 5 | 2

2. Primary Outcome: Incidence of Laboratory Abnormalities
Description: Number (count) of participants that experienced a Grade 3 or higher laboratory toxicity (hematology and chemistry). Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), v4.03. Grade 1 = mild, no intervention needed; Grade 2 = moderate, minimal intervention needed; Grade 3 = severe or medically significant, hospitalization is required; Grade 4 = life-threatening, urgent intervention needed; Grade 5 = death related to adverse event.
Time Frame: Approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant)
Number analyzed (Participants) | 6 | 8
Participants
  Any chemistry test | 4 | 3
  Amylase (iu/l) | 3 | 0
  Alanine aminotransferase (iu/l) | 1 | 1
  Aspartate aminotransferase (iu/l) | 1 | 0
  Total bilirubin (mg/dl) | 3 | 0
  Uric acid (mg/dl) | 1 | 0
  Lipase (iu/l) | 0 | 1
  Sodium (meq/l) | 0 | 1
  Any hematology test | 6 | 5
  Hemoglobin (g/dl) | 3 | 0
  Lymphocytes (x10^3/ul) | 6 | 1
  Neutrophils (x10^3/ul) | 6 | 4
  Platlets (x10^3/ul) | 6 | 4
  White blood cell count (x10^3/ul) | 6 | 5

3. Primary Outcome: 1-year Survival Rate
Description: 1-year survival rate estimated using Kaplan-Meier methods The start date for overall survival is the day of alloSCT.
Time Frame: 12 months
Population: All treated patients set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant)
Number analyzed (Participants) | 6 | 8
percentage of participants | 0 [NA to NA] — Insufficient participants with events to calculate confidence interval. | 75 [31 to 93]

4. Primary Outcome: Rate of MRD Negativity
Description: Rate of MRD (minimal residual disease) negativity at Day -1 (1 day prior to transplant) and Day 30 post-transplant (Part A only)
Time Frame: 30 days
Population: All treated patients set, pre-allo cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pre-allo (Before Stem Cell Transplant)
Number analyzed (Participants) | 6
Percentage of participants
  Day -1 Rate of MRD Negativity | NA [NA to NA] — Insufficient number of participants with events to estimate rate
  Day 30 Rate of MRD Negativity | 75 [19.4 to 99.4]

5. Secondary Outcome: Best Response of CR or CRi
Description: Percentage of patients who achieved a best response of CRi (complete remission with incomplete blood count recovery) or CR (complete remission)
Time Frame: 9 weeks
Population: Part A (pre-alloSCT) only
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-allo (Before Stem Cell Transplant)
Number analyzed (Participants) | 6
Participants | 4

6. Secondary Outcome: Duration of Response
Description: Defined as the time from the start of the first documented complete response (CR) or complete remission with incomplete blood count recovery (CRi) to the documentation of relapse or death due to any cause.
Time Frame: 9 weeks
Population: Part A (pre-alloSCT) only
Measure: Median (Full Range); unit: weeks
Arm/Group | Pre-allo (Before Stem Cell Transplant)
Number analyzed (Participants) | 6
weeks | 6.57 [3 to 9]

7. Secondary Outcome: Overall Survival
Description: Defined as the time from the day of alloSCT to the date of death due to any cause.
Time Frame: Approximately 96 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant)
Number analyzed (Participants) | 6 | 8
weeks | 11.07 [7.43 to 15.71] | NA [31.14 to NA] — <50% of participants experienced an event

ADVERSE EVENTS:
Time Frame: Up to approximately 1 year
Description: Treatment-emergent adverse events: a newly occurring or worsening adverse event after the first dose of study drug.
Arm/Group | Pre-allo (Before Stem Cell Transplant) | Post-allo (After Stem Cell Transplant)
All-Cause Mortality (participants affected / at risk) | 6/6 | 2/8
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-allo (Before Stem Cell Transplant) (N=6) | Post-allo (After Stem Cell Transplant) (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0
Graft versus host disease in lung (Immune system disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Venoocclusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-allo (Before Stem Cell Transplant) (N=6) | Post-allo (After Stem Cell Transplant) (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 2 | 0
Face oedema (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 4
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 5 | 1
Pyrexia (General disorders) | 1 | 1
Graft versus host disease in eye (Immune system disorders) | 0 | 1
Candida infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Respirovirus test positive (Investigations) | 0 | 1
Staphylococcus test positive (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Memory impairment (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Bladder hypertrophy (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery wall hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
No patients were enrolled in Phase 2 due to study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02614560/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02614560/SAP_001.pdf